CLINICAL TRIAL: NCT03663049
Title: Trial of Statin Holiday in Patients Receiving Maintenance Dialysis
Brief Title: The Impact of Statin Holiday in Dialysis Patients Over 70 Years Old on Mental Function, Physical Function and Frailty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Julia Schneider, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 210890
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: ESRD; Cardiovascular Diseases
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Two arms in the study. Patients will be randomized to either continue medication in the statin group or discontinue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): These patients will continue as statins as usual.
- Discontinue statin (Experimental): Patients randomized to this group will stop using the statins they are currently prescribed and will not use their statin medication for 12 weeks.
  Interventions: Drug: discontinue statin

INTERVENTIONS:
Drug: discontinue statin — Discontinue statin as prescribed for 12 weeks
  Arms: Discontinue statin

SUMMARY:
Patients who are on chronic dialysis and 70 and older are frequently on multiple medications including statins. However, the benefit of statins in dialysis patient population is uncertain. Several randomized trials showed no benefit of statins on mortality in dialysis patient population. Guidelines recommend not starting statins in patients on dialysis who are not already taking them. However, there are no guidelines on what to do in patients who are already taking statins. The investigators are doing a short pilot study to discontinue statin in our dialysis patient population and evaluating the effects on discontinuation of statins on quality of life, cognition, as physical strength.

DETAILED DESCRIPTION:
Dialysis patients who are 70 years and older suffer from cognitive dysfunction, physical impairment, and frailty. Polypharmacy in this subgroup of patients is prevalent and can lead to drug toxicities and increased side effects which can contribute to adverse outcomes such as worsening cognitive decline and increased frailty. One frequent component of polypharmacy in dialysis patient population is the use of statins. The use of statins, however, has not been proven to be beneficial in this patient population. While statin medications have been shown to reduce atherosclerotic cardiovascular disease in adults without dialysis dependent chronic kidney disease (CKD), the benefit of statin use in chronic dialysis patients has not been proven. A Cochrane meta-analysis published in 2013 included 25 trials of statin medications in patients receiving maintenance dialysis (total of 8289 patients) and found no benefit of statin medications for preventing atherosclerotic cardiovascular disease events or mortality. The meta-analysis did note that evidence for side effects for statins was incomplete and potential harms from statin medications remain uncertain in this population. Furthermore, statins have recently come under scrutiny by the FDA with regards to their safety due to associations with memory loss and weakness.

Previous clinical trials of statins only assessed the known adverse effects of statins such as abnormal liver function tests and acute kidney injury, adverse effects that occur rarely (< 1%). Trials did not assess other side effects such as cognitive decline or muscle weakness that may be more common in older patients with kidney failure. The aim of this pilot study is to examine the potential side effects of statin medication use in older patients receiving dialysis by conducting a randomized pilot trial of a statin holiday (3 months of discontinuation) vs. no holiday and measuring changes in cognitive function, muscle strength, quality of life and frailty. The investigators hypothesize that measures of cognitive function, grip strength, quality of life and overall frailty will improve after 6 weeks of discontinuation of statins. After obtaining informed consent, patients will complete assessments of quality of life (SF-20), cognition, muscle strength and frailty at baseline and again at 6 and 12 weeks after statin holiday (intervention group) vs. no statin holiday (control group). All patients will resume statin medications after the 3 month trial. The overall goal is to determine whether changes in cognition, strength, frailty or quality of life can be measured using standard instruments. If changes can be detected, pilot data from this study will be used to design a larger trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 70 years and older,
2. Receiving maintenance dialysis for at least 6 months,
3. Must be on a statin medication,
4. Receiving dialysis at the Loyola University Medical Center dialysis unit ,
5. Can be on hemodialysis or peritoneal dialysis,

Exclusion Criteria:

1. Age less than 70 years old
2. Any recent hospital admission (within 2 weeks)
3. Recent dialysis start (within 6 months)
4. Any cancer diagnosis, with exception of innocuous skin cancers and previously treated cancers
5. Any recent (< 1 year) solid organ transplant
6. Active on kidney transplant wait list
7. Recent acute coronary event (e.g. recent NSTEMI, stent, angioplasty, CABG) within 6 months
8. Non-English speaking
9. Diagnosis of dementia
10. Patients who are unable to provide informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | Change in quality of life over 12 weeks
  Change in quality of life will be measured by the Short Form Survey 20 (SF-20). The survey assesses quality of life via 20 questions across 6 domains: physical functioning (6 questions), role functioning (2 questions), social functioning (1 question), mental health (5 questions), health perceptions (5 questions), and pain (1 question). Scores across each of these domains are reported on a 0% to 100% scale, with 0% representing the worst possible score in that domain and 100% the best possible score.

SECONDARY OUTCOMES:
Change in handgrip strength | Change in handgrip strength over 12 weeks
  Handgrip strength will be measured at baseline and again at 6 and 12 weeks

OTHER OUTCOMES:
Change in cognition | Change in cognition over 12 weeks
  Cognition will be measured with trail making test at baseline and again at 6 and 12 weeks
Change in frailty | Change in frailty at 12 weeks
  Frailty will be measured with the Fatigue, Resistance, Aeorbic, Illnesses, and Loss of weight (FRAIL) questionnaire at baseline and again at 6 and 12 weeks. The questionnaire rates each of the five items as 0 for no and 1 for yes, with a total score of 5 possible. Scoring scale: 1-2= pre-frail; 3 or greater=frailty
Change in mobility | Change in mobility at 12 weeks
  Fall risk will be measured with the Get up and go test at baseline and again at 6 and 12 weeks. Time interpretation scale: 10 seconds or less=normal; 20 seconds or less= good mobility; 20 seconds or more = mobility problems, need for a mobility aid

CONTACTS AND LOCATIONS:
Overall Officials: Julia Schneider, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark DA, Khan U, Kiberd BA, Turner CC, Dixon A, Landry D, Moffatt HC, Moorhouse PA, Tennankore KK. Frailty in end-stage renal disease: comparing patient, caregiver, and clinician perspectives. BMC Nephrol. 2017 May 2;18(1):148. doi: 10.1186/s12882-017-0558-x. PMID 28464924
- [Background] McIntyre C, McQuillan R, Bell C, Battistella M. Targeted Deprescribing in an Outpatient Hemodialysis Unit: A Quality Improvement Study to Decrease Polypharmacy. Am J Kidney Dis. 2017 Nov;70(5):611-618. doi: 10.1053/j.ajkd.2017.02.374. Epub 2017 Apr 14. PMID 28416321
- [Background] St Peter WL. Management of Polypharmacy in Dialysis Patients. Semin Dial. 2015 Jul-Aug;28(4):427-32. doi: 10.1111/sdi.12377. Epub 2015 Apr 9. PMID 25864928
- [Background] Fellstrom BC, Jardine AG, Schmieder RE, Holdaas H, Bannister K, Beutler J, Chae DW, Chevaile A, Cobbe SM, Gronhagen-Riska C, De Lima JJ, Lins R, Mayer G, McMahon AW, Parving HH, Remuzzi G, Samuelsson O, Sonkodi S, Sci D, Suleymanlar G, Tsakiris D, Tesar V, Todorov V, Wiecek A, Wuthrich RP, Gottlow M, Johnsson E, Zannad F; AURORA Study Group. Rosuvastatin and cardiovascular events in patients undergoing hemodialysis. N Engl J Med. 2009 Apr 2;360(14):1395-407. doi: 10.1056/NEJMoa0810177. Epub 2009 Mar 30. PMID 19332456
- [Background] Holdaas H, Holme I, Schmieder RE, Jardine AG, Zannad F, Norby GE, Fellstrom BC; AURORA study group. Rosuvastatin in diabetic hemodialysis patients. J Am Soc Nephrol. 2011 Jul;22(7):1335-41. doi: 10.1681/ASN.2010090987. Epub 2011 May 12. PMID 21566054
- [Background] Baigent C, Landray MJ, Reith C, Emberson J, Wheeler DC, Tomson C, Wanner C, Krane V, Cass A, Craig J, Neal B, Jiang L, Hooi LS, Levin A, Agodoa L, Gaziano M, Kasiske B, Walker R, Massy ZA, Feldt-Rasmussen B, Krairittichai U, Ophascharoensuk V, Fellstrom B, Holdaas H, Tesar V, Wiecek A, Grobbee D, de Zeeuw D, Gronhagen-Riska C, Dasgupta T, Lewis D, Herrington W, Mafham M, Majoni W, Wallendszus K, Grimm R, Pedersen T, Tobert J, Armitage J, Baxter A, Bray C, Chen Y, Chen Z, Hill M, Knott C, Parish S, Simpson D, Sleight P, Young A, Collins R; SHARP Investigators. The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. Lancet. 2011 Jun 25;377(9784):2181-92. doi: 10.1016/S0140-6736(11)60739-3. Epub 2011 Jun 12. PMID 21663949
- [Background] Olyaei A, Steffl JL, MacLaughlan J, Trabolsi M, Quadri SP, Abbasi I, Lerma E. HMG-CoA reductase inhibitors in chronic kidney disease. Am J Cardiovasc Drugs. 2013 Dec;13(6):385-98. doi: 10.1007/s40256-013-0041-4. PMID 23975627
- [Background] Wanner C, Tonelli M; Kidney Disease: Improving Global Outcomes Lipid Guideline Development Work Group Members. KDIGO Clinical Practice Guideline for Lipid Management in CKD: summary of recommendation statements and clinical approach to the patient. Kidney Int. 2014 Jun;85(6):1303-9. doi: 10.1038/ki.2014.31. Epub 2014 Feb 19. PMID 24552851
- [Background] Manley HJ, McClaran ML, Overbay DK, Wright MA, Reid GM, Bender WL, Neufeld TK, Hebbar S, Muther RS. Factors associated with medication-related problems in ambulatory hemodialysis patients. Am J Kidney Dis. 2003 Feb;41(2):386-93. doi: 10.1053/ajkd.2003.50048. PMID 12552501
- [Background] Talar Markossian, Holly Kramer, Nicholas Burge, et a. Utilization of statins in U.S. Veterans with dialysis-dependent chronic kidney disease. Health Sciences Research. 2018 Under review
- [Background] Kurella Tamura M, Larive B, Unruh ML, Stokes JB, Nissenson A, Mehta RL, Chertow GM; Frequent Hemodialysis Network Trial Group. Prevalence and correlates of cognitive impairment in hemodialysis patients: the Frequent Hemodialysis Network trials. Clin J Am Soc Nephrol. 2010 Aug;5(8):1429-38. doi: 10.2215/CJN.01090210. Epub 2010 Jun 24. PMID 20576825
- [Background] Johansen KL, Chertow GM, Jin C, Kutner NG. Significance of frailty among dialysis patients. J Am Soc Nephrol. 2007 Nov;18(11):2960-7. doi: 10.1681/ASN.2007020221. Epub 2007 Oct 17. No abstract available. PMID 17942958
- [Background] Herzog CA, Asinger RW, Berger AK, Charytan DM, Diez J, Hart RG, Eckardt KU, Kasiske BL, McCullough PA, Passman RS, DeLoach SS, Pun PH, Ritz E. Cardiovascular disease in chronic kidney disease. A clinical update from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2011 Sep;80(6):572-86. doi: 10.1038/ki.2011.223. Epub 2011 Jul 13. PMID 21750584
- [Background] Isoyama N, Qureshi AR, Avesani CM, Lindholm B, Barany P, Heimburger O, Cederholm T, Stenvinkel P, Carrero JJ. Comparative associations of muscle mass and muscle strength with mortality in dialysis patients. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1720-8. doi: 10.2215/CJN.10261013. Epub 2014 Jul 29. PMID 25074839
- [Background] Dong J, Pi HC, Xiong ZY, Liao JL, Hao L, Liu GL, Ren YP, Wang Q, Duan LP, Zheng ZX. Depression and Cognitive Impairment in Peritoneal Dialysis: A Multicenter Cross-sectional Study. Am J Kidney Dis. 2016 Jan;67(1):111-8. doi: 10.1053/j.ajkd.2015.06.025. Epub 2015 Aug 6. PMID 26255306
- [Background] Fazekas G, Fazekas F, Schmidt R, Kapeller P, Offenbacher H, Krejs GJ. Brain MRI findings and cognitive impairment in patients undergoing chronic hemodialysis treatment. J Neurol Sci. 1995 Dec;134(1-2):83-8. doi: 10.1016/0022-510x(95)00226-7. PMID 8747848
- [Background] Sehgal AR, Grey SF, DeOreo PB, Whitehouse PJ. Prevalence, recognition, and implications of mental impairment among hemodialysis patients. Am J Kidney Dis. 1997 Jul;30(1):41-9. doi: 10.1016/s0272-6386(97)90563-1. PMID 9214400
- [Background] Lopes AA, Lantz B, Morgenstern H, Wang M, Bieber BA, Gillespie BW, Li Y, Painter P, Jacobson SH, Rayner HC, Mapes DL, Vanholder RC, Hasegawa T, Robinson BM, Pisoni RL. Associations of self-reported physical activity types and levels with quality of life, depression symptoms, and mortality in hemodialysis patients: the DOPPS. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1702-12. doi: 10.2215/CJN.12371213. Epub 2014 Oct 2. PMID 25278548
- [Background] Topolski TD, LoGerfo J, Patrick DL, Williams B, Walwick J, Patrick MB. The Rapid Assessment of Physical Activity (RAPA) among older adults. Prev Chronic Dis. 2006 Oct;3(4):A118. Epub 2006 Sep 15. PMID 16978493
- [Background] Painter P, Marcus RL. Assessing physical function and physical activity in patients with CKD. Clin J Am Soc Nephrol. 2013 May;8(5):861-72. doi: 10.2215/CJN.06590712. Epub 2012 Dec 6. PMID 23220421
- See also: Drug Safety and Availability - FDA Drug Safety Communication: Important safety label changes to cholesterol-lowering statin drugs [Internet].: Center for Drug Evaluation and Research [cited Mar 9, 2018] — http://www.fda.gov/Drugs/DrugSafety/ucm293101.htm